CLINICAL TRIAL: NCT01254591
Title: Tumor Angiogenesis in Non-Small Cell Lung (NSCLC), Colorectal, Breast, Esophageal, Head and Neck Cancer: Radiology-Pathology and Prognostic Correlation
Brief Title: Positron Emission Tomography/Computed Tomography Scanning Before Surgery in Patients With Non-Small Cell Lung Cancer, Colorectal Cancer, Breast Cancer, Esophageal Cancer, or Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London (UCL) Cancer Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000689973; UCL-TUMOR-ANGIOGENESIS; EU-21086
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Esophageal Cancer; Head and Neck Cancer; Lung Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer; stage IIIA colon cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage I hypopharyngeal cancer; stage II hypopharyngeal cancer; stage III hypopharyngeal cancer; stage I laryngeal cancer; stage II laryngeal cancer; stage III laryngeal cancer; stage I lip and oral cavity cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer; stage I nasopharyngeal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage I oropharyngeal cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer; stage I paranasal sinus and nasal cavity cancer; stage II paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; tongue cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — fluoromisonidazole; Magnetic Resonance Spectroscopy; 5-fluoropentyl-2-methylmalonic acid; Fluorodeoxyglucose F18; Rubidium-82

INTERVENTIONS:
Other: 18F-fluoromisonidazole
Other: fluorescence angiography
Other: laboratory biomarker analysis
Procedure: infrared thermography
Procedure: magnetic resonance imaging
Procedure: therapeutic conventional surgery
Radiation: [18F]-ML-10
Radiation: fludeoxyglucose F 18
Radiation: rubidium Rb-82

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography/computed tomography (PET/CT) scanning before surgery, may help measure the extent of disease.

PURPOSE: This clinical trial is studying PET/CT scanning before surgery in patients with non-small cell lung cancer, colorectal cancer, breast cancer, esophageal cancer, or head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the ability of preoperative fludeoxyglucose F 18 positron emission tomography/computed tomography (PET/CT) scanning in assessing tumor angiogenesis in patients with potentially operable non-small cell lung cancer, colorectal cancer, breast cancer, esophageal cancer, or head and neck cancer.
* To determine the ability of preoperative fludeoxyglucose F 18 PET/CT scanning in assessing prognosis by means of measuring angiogenesis in these patients.

OUTLINE: All patients undergo fludeoxyglucose F 18 positron emission tomography/computed tomography (PET/CT) scanning for staging, tumor perfusion measurement/angiogenesis, and glucose metabolism. If staging confirms operable disease, then the patient proceeds to surgery as planned. Resected tumor tissue samples are examined for tumor angiogenesis in the various cancer types.

Some patients undergo a half-dose of rubidium Rb-82 or 18F-fluoromisonidazole or [18F]-ML-10 PET scan or fluorescence angiography. Patients with colorectal cancer undergo a CT scan for perfusion of the tumor after the staging PET/CT. Patients with breast cancer undergo infrared thermometry as well as a MRI scan for staging and to predict angiogenesis.

After completion of study therapy, patients are followed up at 1 month and then every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer, colorectal cancer, breast cancer, esophageal cancer, or head and neck cancer

  * Potentially operable disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Not specified
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-11; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Clinical, radiological, and pathological correlation
Prognosis (6-month, 1-year, 3-year, and 5-year mortality including local/distance recurrence rates)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ell, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital, London, England, United Kingdom